CLINICAL TRIAL: NCT02049580
Title: Multi-center, Phase II Study to Assess the Safety and Efficacy of Haploidentical Bone Marrow Transplantation Using Reduced Intensity Conditioning(RIC)Regimen and Post-transplant Cyclophosphamide,in Patients With Poor Prognosis Lymphomas
Brief Title: Reduced Intensity Conditioning (RIC) Regimen and Post-transplant Cyclophosphamide in Haploidentical Bone Marrow Transplantation in in Patients With Poor Prognosis Lymphomas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2011-005
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Lymphoma
Keywords: lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Thiotepa; fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RIC regimen (Experimental): Thiotepa, Fludarabine, Cyclophosphamide pre- and post- transplantation.
  Interventions: Drug: Thiotepa; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Thiotepa — Thiotepa (10 mg/kg /day) will be administered every 12 h, at day -6
  Other Names: Tepadina
Drug: Fludarabine — Fludarabine (30mg/m2/day x 4 days) will be dosed according to renal function. For decreased creatinine clearance (CCr) (≤ 61 mL/min) Fludarabine dosage should be reduced as follows:
  CCr 46-60 mL/min, fludarabine = 24 mg/ m2/day
  Other Names: Fludara
Drug: Cyclophosphamide — Pre-transplantation Cyclophosphamide(Cy) 30 mg/kg/day will be administered as a 1-2 hour intravenous infusion with a high volume fluid flush on Days -5.
  Cy will be dosed according to the recipient's ideal body weight (IBW), unless the patient weighs more than 125% of IBW, in which case the drug will be dosed according to the Adjusted IBW (AIBW)
  Cyclophosphamide [50 mg/kg/day IBW] will be given on Day 3 post-transplant (between 60 and 72 hours after marrow infusion) and on Day 4 post-transplant (approximately 24 hours after Day 3 cyclophosphamide). Cyclophosphamide will be given as an IV infusion over 1-2 hours (depending on volume).
  Other Names: Endoxan

SUMMARY:
Study to test feasibility and efficacy of T-replete Bone Marrow (BM), infused after a RIC regimen and post-transplantation Cyclophosphamide (Cy), in patients with poor prognosis lymphomas.

DETAILED DESCRIPTION:
Allogeneic stem cell transplantation (ALLO) is the treatment of choice for many hematological diseases. However, HLA identical donor (sibling or unrelated) is available for 50-60% of patients and alternative donors are needed. Haploidentical donors have been used for many years, mostly after extensive T-cell depletion of peripheral stem cell, to avoid Graft Versus Host Disease (GVHD). Recently, promising data have been reported with haploidentical transplantation using T-replete bone marrow (BM) and high-dose cyclophosphamide (Cy) post-transplantation. However, the conditioning regimen did not contain drugs active against hemopathies, enhancing the relapse risk.

In this study, the investigators want to test the feasibility and efficacy of T-replete BM, infused after a RIC regimen and post-transplantation Cy, in patients with poor prognosis lymphoproliferative diseases.

The RIC regimen consisted of modified regimen used in different studies conducted in Italy on behalf GITMO.

ELIGIBILITY:
* Signed and dated IEC-approved informed consent
* Age ≥ 18-70 years old.
* Performance Status Karnofsky ≥ 80% (see appendix B)
* HLA typing will be performed at high resolution (allele level) for the HLA-A, HLA -B, HLA Cw, HLA-DRB1, and HLA-DQB1 loci. A minimum match of 5/10 is required. An unrelated donor search is not required for a patient to be eligible for this protocol if the clinical situation dictates an urgent transplant.
* The donor and recipient must be identical, as determined by high resolution typing, at least one allele of each of the following genetic loci: HLA-A, HLA-B, HLA-Cw, HLA-DRB1, and HLA-DQB1.
* Patients with lymphoma (any histology) relapsed after high dose chemotherapy and in partial remission, complete remission or stable disease after the last CT line.

  1. Hodgkin's lymphoma: Patients refractory to at least 2 CT lines, and included in tandem auto-allo program
  2. Diffuse large B cell lymphoma: Refractory to second line salvage chemotherapy (patients in partial remission, stable disease or progressive). These patients have to be in partial remission, complete remission or stable disease after one o more further CT line.
  3. Peripheral T cell lymphoma: Patients failing to achieve a complete remission after first line CT.
  4. Low grade lymphomas (follicular and non follicular: Patients refractory to rituximab containing regimens. Patients relapsing after at least 2 lines CT. The duration of remission should be < 1 year.
  5. Chronic lymphatic leukemia: Patients with refractory or relapsing (response duration < 1 year) disease after R-Fludarabine CT
  6. Mantle cell lymphoma: Patients relapsing or refractory after first line conventional CT.
* Absence of HLA identical sibling and 10/10 unrelated donor
* Patients with adequate physical function as measured by:

Cardiac: Left ventricular ejection fraction at rest must be ≥ 40% Hepatic: Bilirubin ≤ 2.5 mg/dL; and ALT, AST, and Alkaline Phosphatase ≤ 5 x ULN.

Renal: Creatinine clearance or GFR ≥ 50 mL/min/1.73 m2. Pulmonary: FEV1, FVC, DLCO ≥ 50% predicted (corrected for hemoglobin); if unable to perform pulmonary function tests, then O2 saturation ≥ 92% on room air.

Exclusion Criteria:

* Presence of HLA-matched, related donor (HLA-A, -B, -DRB1)
* Presence of matched unrelated donor (10/10), available on time.
* Pregnancy or breast-feeding.
* Evidence of HIV infection or known HIV positive serology.
* Current uncontrolled bacterial, viral or fungal infection
* Evidence of progression of clinical symptoms or radiologic findings.
* Prior allogeneic hematopoietic stem cell transplant.
* Central Nervous System (CNS) lymphoma localization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-08 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Procedure activity | 1 year
  1-year Progression Free Survival (PFS) to evaluate the activity of the procedure (taking into account an excess of toxicity). It is assumed that at 1-year a proportion of patients progression free of 20% or lower will be considered to be clinically unworthy, whereas a proportion of 40% or higher will be assumed to be of potential interest.

SECONDARY OUTCOMES:
Neutrophils recovery | 1 year
  Neutrophils will be measured at different time points of increasing lenght up to 1 year after transplant and then if clinically indicated
Platelets recovery | 1 year
  Platelets will be measured at different time points of increasing lenght up to 1 year after transplant and then if clinically indicated
Incidence of graft failure | 1 year
Cumulative incidence of acute and chronic GVHD | 1 year
Incidence of infections | 1 year
  Possible infections will be monitored for a time period of 1 year post-transplantation and then if clinically required
Cumulative incidence of relapse/progression | 1 year
Treatment related mortality (TRM) | 1 year
Immunological reconstitution | 1 year
  T, B and NK subsets will be analysed in deep using cytofluorimetry and functional tests.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Castagna, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, MI, Italy

REFERENCES:
- [Derived] Roberto A, Castagna L, Zanon V, Bramanti S, Crocchiolo R, McLaren JE, Gandolfi S, Tentorio P, Sarina B, Timofeeva I, Santoro A, Carlo-Stella C, Bruno B, Carniti C, Corradini P, Gostick E, Ladell K, Price DA, Roederer M, Mavilio D, Lugli E. Role of naive-derived T memory stem cells in T-cell reconstitution following allogeneic transplantation. Blood. 2015 Apr 30;125(18):2855-64. doi: 10.1182/blood-2014-11-608406. Epub 2015 Mar 5. PMID 25742699